CLINICAL TRIAL: NCT06955507
Title: Effect of Foot Reflexology on Perineal Pain, Fatigue and Healing Quality in Primiparous Patients Undergoing Episiotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Neziha Bayazıt, MIDWIFE, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSU-EBE-NB-01
Record Dates: First submitted 2025-01-30; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: Episiotomy
Keywords: Birth; reflexology; perineal pain; fatigue; quality of recovery
MeSH Terms: conditions — Fatigue | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Two groups will be created as experimental and control groups among primiparous women who have undergone episiotomy.
Masking Description: Two groups will be created as experimental and control groups among primiparous women who have undergone episiotomy, and reflexology will be applied to the women in the experimental group and will not be applied to the other group. Necessary questionnaires will be filled out in the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group to apply foot reflexology technique to primiparas who underwent episiotomy (Experimental): First Measurement: Personal Information Form, VAS and YİGBÖ will be applied 3 hours after birth. Then, the first foot reflexology lasting on average 30 minutes will be applied to these women.
  Second Measurement: Immediately after the first foot reflexology, the pain intensity will be re-evaluated with VAS.
  Third Measurement: 15 hours after birth, the pain level will be re-evaluated with VAS and then the experimental group will be applied a second foot reflexology lasting on average 30 minutes.
  Fourth Measurement: VAS and YİGBÖ will be applied immediately after the second foot reflexology.
  Fifth Measurement: DSİKÖ will be filled in at the 24th hour.
  Interventions: Behavioral: reflexology
- Not Applying Foot Reflexology to Primiparous Women Who Underwent Episiotomy (No Intervention): First Measurement: Personal Information Form, VAS and YİGBÖ will be applied 3 hours after birth.
  Second Measurement: Pain intensity will be re-evaluated with VAS immediately after the first foot reflexology simultaneously with the foot reflexology application chart applied to the experimental group.
  Third Measurement: Pain level will be re-evaluated with VAS 15 hours after birth.
  Fourth Measurement: VAS and YİGBÖ will be applied simultaneously with the foot reflexology application chart applied to the experimental group and immediately after the second foot reflexology.
  Fifth Measurement: DSİKÖ will be filled out at the 24th hour before discharge.

INTERVENTIONS:
Behavioral: reflexology — Foot reflexology will be applied by the researcher Neziha BAYAZIT, who will receive training on this subject, in the quietest and most comfortable position possible. Foot reflexology will be applied by the researcher to the women in the experimental group. The researcher will receive training on foot reflexology before the study. In the clinic where the study will be conducted, the hours of foot reflexology application will be determined considering the analgesic treatment protocol applied. Accordingly, analgesic treatment is routinely applied to the women who will receive foot reflexology at the 4th hour according to hospital procedure. Foot reflexology will be applied by the researcher at least 1 hour before the analgesic treatment (3rd hour - 15th hour after birth). The same foot reflexology will be repeated 12 hours later at the 15th hour after the first foot reflexology is performed at the 3rd hour after birth. Each woman will be given an explanation before the application. Foot r
  Arms: Experimental group to apply foot reflexology technique to primiparas who underwent episiotomy

SUMMARY:
The act of giving birth can expose women to many risks during pregnancy and the birth process. It causes long-term emotional problems in pregnant women who experience labor pain and negatively affects their mental health. Episiotomy is a method applied to facilitate the birth of the baby by enlarging the vaginal opening. The postpartum period can significantly affect the lives of every mother, especially mothers who have had an episiotomy and vaginal birth. Many factors such as pain, fatigue and the negative effects of anesthetic drugs can negatively affect postpartum comfort and breastfeeding, causing late mother-baby bonding. With the support and information given to women during this period, women can be helped to make healthier and more accurate choices. They increasingly prefer natural methods to cope with problems that arise after birth. Some methods are used to accelerate recovery and prevent potential problems. Reflexology is an energy balancing system and special pressure method applied to reflex points with rubbing, squeezing and patting movements to increase rapid recovery.

DETAILED DESCRIPTION:
The researcher will apply the face-to-face interview method to women who have undergone episiotomy in the postpartum ward located within the additional service building of Kahramanmaraş Necip Fazıl City Hospital, Maternity and Child.

Experimental Group;

First Measurement: Personal Information Form, VAS and YİGBÖ will be applied 3 hours after birth. Then, the first foot reflexology lasting on average 30 minutes will be applied to these women.

Second Measurement: Immediately after the first foot reflexology, the pain intensity will be re-evaluated with VAS.

Third Measurement: 15 hours after birth, the pain level will be re-evaluated with VAS and then the experimental group will be applied foot reflexology for a second time lasting on average 30 minutes.

Fourth Measurement: VAS and YİGBÖ will be applied immediately after the second foot reflexology.

Fifth Measurement: DSİKÖ will be filled in at the 24th hour.

Control Group; First Measurement: Personal Information Form, VAS and YİGBÖ will be applied 3 hours after birth.

Second Measurement: The pain intensity will be re-evaluated with VAS immediately after the first foot reflexology simultaneously with the foot reflexology application schedule applied to the experimental group.

Third Measurement: The pain level will be re-evaluated with VAS 15 hours after birth.

Fourth Measurement: VAS and YİGBÖ will be applied immediately after the second foot reflexology simultaneously with the foot reflexology application schedule applied to the experimental group.

Fifth Measurement: DSİKÖ will be filled in before discharge at the 24th hour. Foot Reflexology Application Procedure Foot reflexology will be applied by the researcher Neziha BAYAZIT, who will receive training on this subject, in the quietest and most comfortable position possible. Foot reflexology will be applied to the women in the experimental group by the researcher. The researcher will receive training on foot reflexology before the study. In the clinic where the study will be conducted, the foot reflexology application hours will be determined considering the analgesic treatment protocol applied. Accordingly, analgesic treatment is routinely applied to women who will receive foot reflexology at the 4th hour according to hospital procedure. Foot reflexology will be applied by the researcher at least 1 hour before the procedure analgesic treatment (3-15 hours after birth). The first foot reflexology will be applied at 3 hours after birth and the same foot reflexology will be repeated 12 hours later at 15 hours. Each woman will be given an explanation before the application. Foot reflexology will be applied in the patient rooms. The application will take approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Being literate,
* Having a gestational age of 37-42 weeks,
* Having a newborn weighing between 2500-4000 grams,
* Expressing that perineal pain is "moderate" or "severe",
* Being open to communication.

Exclusion Criteria:

* No other lacerations (anal sphincter injury, 3rd degree perineal laceration) other than episiotomy,
* Newborn weighing between 2500-4000 grams,
* Perineal pain stated as "moderate" or "severe",
* No complications related to mother and baby in the postpartum period (bleeding, hypertension, babies taken to neonatal intensive care unit, etc.),
* No cognitive problems,
* No conditions that make reflexology application undesirable such as thrombophlebitis, deep vein thrombosis, epilepsy, febrile illnesses, etc.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Our study consists of women who gave birth for the first time.
Enrollment: 68 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Effect of Foot Reflexology on Perineal Pain, Fatigue and Quality of Recovery in Primiparous Women Undergoing Episiotomy | up to 24. hours after birth
  In primiparas who underwent episiotomy, the experimental group was the group to which foot reflexology was applied, while the control group was the group to which foot reflexology was not applied. A personal information form, Visual Analog Scale and Visual Similarity Scale for Fatigue will be filled out for both groups. The VAS is numbered from 0 to 10. Findings have shown that VAS ratings of 0 to 4 mm per 100 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain. Scale ratings assess the effect of foot reflexology on episiotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Necip Fazıl Hospital Maternity and Child Additional Service Building, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)